CLINICAL TRIAL: NCT03711422
Title: A Dose Finding Study of Continuous and Intermittent High-dose (HDI) Afatinib (EGFR TKI) on CNS Metastases and Leptomeningeal Disease (LMD) in Patients With Advanced Refractory EGFR Mutation Positive Non-small Cell Lung Cancer
Brief Title: Afatinib on CNS Metastases and LMD in EGFR Mutation Positive NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to close the trial made due to low recruitment.
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.275
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2021-04

CONDITIONS: Non-small Cell Lung Cancer; Leptomeningeal Disease; Central Nervous System Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Standard dose oral afatinib. If patients in Part A do not benefit from the regimen, they can be enrolled into Part B
  Interventions: Drug: Afatinib
- Part B (Experimental): Intermittent high dose oral afatinib
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 40mg daily
  Other Names: Gilotrif
  Arms: Part A
Drug: Afatinib — 160mg for 3 days every 3 weeks
  Other Names: Gilotrif
  Arms: Part B

SUMMARY:
Brain metastases occurs in up to 50% of patients with EGFR mutant NSCLC. Leptomeningeal disease is a subset of patients with brain metastases for which there remains an unmet need. This trial aims to evaluate the role of two dosing schedules of afatinib in management of leptomeningeal disease in EGFR mutant NSCLC, specifically to determine Central Nervous System (CNS) penetration of afatinib, as well as clinical activity. Patients will start on daily dosing initially followed by pulsed intermittent dosing should we observe no clinical activity. A secondary objective is to identify the resistance spectrum in leptomeningeal disease. It is anticipated that optimal dosing schedule of afatinib e.g. pulsed dosing may improve CNS disease control.

ELIGIBILITY:
Inclusion Criteria:

* Patients progressing locally in the CNS after prior systemic treatment and Whole brain radiotherapy (WBRT)/ Stereotactic radiosurgery (SRS) (or declines radiotherapy), for which no standard therapy options are available
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0-3
* Adequate organ function

  * Absolute neutrophil count (ANC) ≥1500 / mm3 . (ANC >1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the investigator and in discussion with the sponsor).
  * Platelet count ≥75,000 / mm3 .
  * Estimated creatinine clearance > 45ml/min
  * Left ventricular function with resting ejection fraction ≥ 50% or above the institutional Lower Limit of Normal (LLN).
  * Total Bilirubin ≤ 1.5 times upper limit of (institutional/central) normal (Patients with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal)
  * Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ three times the upper limit of (institutional/central) normal (ULN) (if related to liver metastases ≤ five times ULN).
* Written informed consent that is consistent with ICH-GCP guidelines

Exclusion Criteria:

* Symptomatic brain metastases requiring high dose steroids. Patients are excluded from Part A if they develop cerebral manifestation under afatinib. (Those progressing on afatinib will proceed to part B with HDI afatinib)
* Hormonal treatment within 2 weeks prior to start of study treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted) Radiotherapy within 4 weeks prior to randomization, except as follows:

  * Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to randomisation, and
  * Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Known hypersensitivity to afatinib or the excipients of any of the trial drugs
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
* Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly prior to study entry, for the duration of study participation and for at least <XX weeks; 2 weeks for afatinib, XX weeks for comparator,> after treatment has ended.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
* Previous or concomitant malignancies at other sites, except effectively treated nonmelanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Requiring treatment with any of the prohibited concomitant medications listed in Section 4.2.2.1 that cannot be stopped for the duration of trial participation
* Known pre-existing interstitial lung disease
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
* Active hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Afatinib concentration in plasma using standard dosing and high intermittent dosing | Day 1 to Day 29 of drug treatment
  To assess the difference in drug ratio from two difference dosing of afatinib
Afatinib concentration in Cerebral Spinal Fluid (CSF) using standard dosing and high intermittent dosing | Part A: Day 15; Part B: Day 17 and 31
  To assess the difference in drug ratio from two difference dosing of afatinib
Neurological Progression Free Survival | From time of first study drug administration until first occurrence of disease progression, or death from any cause, up to 2 years
Neurological Response Rate | From time of first study drug administration until first occurrence of disease progression, up to 2 years
Overall Survival | From time of first study drug administration to death from any cause, up to 2 years

SECONDARY OUTCOMES:
Cell-free DNA sequencing of Cerebrospinal Fluid | From time of first study drug administration to end of study treatment, up to 2 years
  To detect EGFR T790M and activating mutation status
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 | From time of first study drug administration through to end of study treatment or disease progression, up to 2 years
  To assess the physical, physiological and social functions. The scale ranges from 1="not all all" to 4-"very much"
EORTC Quality of Life Questionnaire Brain Cancer Module | From time of first study drug administration through to end of study treatment or disease progression, up to 2 years
  To assess future uncertainty, visual disorder, motor dysfunction, and communication deficit. The scale ranges from 1="not all all" to 4-"very much"
Incidences of treatment-emergent adverse events (AE) | From time of first study drug administration to 28 days after last treatment administration
  AEs will be graded according to CTCAE, Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffknecht P, Tufman A, Wehler T, Pelzer T, Wiewrodt R, Schutz M, Serke M, Stohlmacher-Williams J, Marten A, Maria Huber R, Dickgreber NJ; Afatinib Compassionate Use Consortium (ACUC). Efficacy of the irreversible ErbB family blocker afatinib in epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI)-pretreated non-small-cell lung cancer patients with brain metastases or leptomeningeal disease. J Thorac Oncol. 2015 Jan;10(1):156-63. doi: 10.1097/JTO.0000000000000380. PMID 25247337
- [Background] Awada AH, Dumez H, Hendlisz A, Wolter P, Besse-Hammer T, Uttenreuther-Fischer M, Stopfer P, Fleischer F, Piccart M, Schoffski P. Phase I study of pulsatile 3-day administration of afatinib (BIBW 2992) in combination with docetaxel in advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):734-41. doi: 10.1007/s10637-012-9880-0. Epub 2012 Nov 17. PMID 23161334